CLINICAL TRIAL: NCT02598115
Title: Impact of the Implementation of Collaborative Pharmaceutical Care on Hospital Admission Drug Prescriptions for Patients 65 Years of Age and Older
Brief Title: Impact of Collaborative Pharmaceutical Care on Hospital Admission Drug Prescriptions for Patients 65 Years of Age and Older
Acronym: MEDREV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PREPS/2014/JMK-01; 2015-A00421-48 (Other: RCB number)
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Aged; Patient Admission; Hospitalization
Keywords: collaborative pharmaceutical care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Before collarborative pharmaceutical care (No Intervention): All clusters start in this arm for 15 days. Following the start of the study, 1 randomly chosen cluster will switch to the experimental arm every 15 days.
  Days 1 to 15: all clusters in the "before arm" Days 16 to 30: 1 cluster in the "Collaborative Pharmaceutical Care" arm Days 31 to 45: 2 clusters in the "Collaborative Pharmaceutical Care" arm Days 46 to 60: 3 clusters in the "Collaborative Pharmaceutical Care" arm Days 61 to 75: 4 clusters in the "Collaborative Pharmaceutical Care" arm Days 76 to 90: 5 clusters in the "Collaborative Pharmaceutical Care" arm Days 91 to 105: all 6 clusters in the "Collaborative Pharmaceutical Care" arm
- After collarborative pharmaceutical care (Experimental): All clusters start in the "No Intervention" arm for 15 days. Following the start of the study, 1 randomly chosen cluster will switch to the experimental arm every 15 days.
  Days 1 to 15: all clusters in the "before arm" Days 16 to 30: 1 cluster in the "Collaborative Pharmaceutical Care" arm Days 31 to 45: 2 clusters in the "Collaborative Pharmaceutical Care" arm Days 46 to 60: 3 clusters in the "Collaborative Pharmaceutical Care" arm Days 61 to 75: 4 clusters in the "Collaborative Pharmaceutical Care" arm Days 76 to 90: 5 clusters in the "Collaborative Pharmaceutical Care" arm Days 91 to 105: all 6 clusters in the "Collaborative Pharmaceutical Care" arm
  Interventions: Other: Collaborative Pharmaceutical Care

INTERVENTIONS:
Other: Collaborative Pharmaceutical Care — The pharmacist performs collaborative pharmaceutical care in the ward: reconciliation of drug treatments and revision of drug prescriptions indicated on the admission drug prescription. He/she emits pharmaceutical interventions recorded on the standardized support provided by the French Society of Clinical Pharmacy. The pharmaceutical interventions are discussed during a collaborative interview.
  Arms: After collarborative pharmaceutical care

SUMMARY:
The primary objective of this study is to evaluate the impact of the implementation of collaborative pharmaceutical care on drug support at admission for patients 65 years of age and older.

This is a cluster-randomized study with a stepped-wedge design. Clusters correspond to participating centers. A randomly selected center is crossed-over into the intervention every fifteen days after the start of inclusions.

DETAILED DESCRIPTION:
The secondary objectives are to evaluate:

A. The potential and observed clinical impact of the implementation of collaborative pharmaceutical care.

B. The acceptance rate of pharmaceutical interventions during collaborative pharmaceutical care.

C. Avoidable costs related to the consumption of care generated by the occurrence of serious adverse drug reactions.

D. The satisfaction of health professionals concerning the transfer of information on the patient's drug therapy carried out as part of collaborative pharmaceutical care.

ELIGIBILITY:
Inclusion Criteria:

* The patient or his/her legal representative was informed about the study
* The patient is admitted as an in-patient to one of the participating hospitals
* The patient is available for 3 months of follow-up

Exclusion Criteria:

* The subject is participating in another drug study
* The subject is under judicial protection
* It is impossible to correctly inform the patient or his/her legal representative
* The patient or his/her legal representative refuses to participate in the study
* The expected life span of the patient is less than the required 3 months of follow-up
* It is impossible to contact the patient after hospitalisation
* Hospitalizatin for longer than 21 days

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 622 (Actual)
Dates: Start 2016-09-19 (Actual); Primary Completion 2016-12-25 (Actual); Study Completion 2016-12-25 (Actual)

PRIMARY OUTCOMES:
Number of patients with at least one preventable medication error | Day 1 (medical prescription at hospital admission)
Number of patients with at least one preventable medication error | Phase 2 (maximum 105 days)
  Number of patients with at least one preventable medication error not accepted by the prescribing doctor during the interventional phase

SECONDARY OUTCOMES:
Preventable medication error rate | Day 1 (medical prescription at hospital admission)
  Potential clinical impact: preventable medication error rate detected in the medical prescription at admission (MPA) according to the level of criticality 1, 2 or 3. This error rate is defined by the ratio of the number of avoidable errors to the number of unrevised lines in the MPA.
Number of patients at high risk for adverse drug events | Day 1 (medical prescription at hospital admission)
  Potential clinical impact: number of patients at high risk for adverse drug events (Trivalle score calculated on the medical prescription at hospital admission)
Readmission rate for in-patient hospitalization | 30 days after hospital discharge (expected maximum of 21 days of hospitalization)
  Clinical impact observed: readmission rate for in-patient hospitalization
Readmission rate for in-patient hospitalization | 90 days after hospital discharge (expected maximum of 21 days of hospitalization)
  Clinical impact observed: readmission rate for in-patient hospitalization
Mortality rate | 30 days after hospital discharge (expected maximum of 21 days of hospitalization)
Mortality rate | 90 days after hospital discharge (expected maximum of 21 days of hospitalization)
Length of hospital stay | hospital discharge (expected maximum of 21 days of hospitalization)
Acceptance rate of pharmaceutical interventions during collaborative interview. | Day 1, hospital admission
Avoided costs related to the occurrence of medication errors (criticality 3) | 90 days after hospital discharge (expected maximum of 21 days of hospitalization)
Satisfaction questionnaire (for health care professionals) on the implementation of collaborative pharmaceutical care | End of study (expected at 195 days)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marie Kinowski, PharmD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (6):
- France (6):
  - CHU de Grenoble - Hôpital Albert Michallon, Grenoble
  - CHU de Nice - Hôpitaux L'Archet 1 et 2, Nice
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes
  - CHU de Rouen - Hôpital Charles Nicolle, Rouen
  - CHRU de Strasbourg - Hôpital de Hautepierre, Strasbourg
  - CHRU de Toulouse - Hôpital Paule de Viguier, Toulouse

REFERENCES:
- [Derived] Leguelinel-Blache G, Bouvet S, Bedouch P, Bachelet B, Chenailler C, Dantin T, Geneletti L, Janes A, Scher F, Cireasa B, Kinowski JM, Castelli C, Roux-Marson C; Working Group "Valorisation of Pharmacist Interventions" of the French Society of Clinical Pharmacy; MEDREV working group. Impact of collaborative pharmaceutical care on older inpatients' medication safety: multicentre stepped-wedge cluster randomised trial (MEDREV Study). BMC Geriatr. 2025 Jul 11;25(1):516. doi: 10.1186/s12877-025-06122-1. PMID 40646458
- [Derived] Leguelinel-Blache G, Castelli C, Roux-Marson C, Bouvet S, Andrieu S, Cestac P, Collomp R, Landais P, Louliere B, Mouchoux C, Varin R, Allenet B; MEDREV Working Group; Bedouch P, Kinowski JM. Impact of collaborative pharmaceutical care on in-patients' medication safety: study protocol for a stepped wedge cluster randomized trial (MEDREV study). Trials. 2018 Jan 8;19(1):19. doi: 10.1186/s13063-017-2412-7. PMID 29310711